CLINICAL TRIAL: NCT00513864
Title: Non-Invasive Assessment of Opioid Analgesia in Children With Sickle Cell Disease
Brief Title: Assessment of Opioid Analgesia in Sickle Cell
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Julia Finkel, MD, Children's National Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3919
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Sickle Cell Disease
Keywords: Opioid Analgesics; Morphine; Codeine; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Dextromethorphan; Codeine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYP2D6- (Active Comparator): This arm consists of subjects that are poor metabolizers (PM) and intermediate metabolizers (IM).
  Interventions: Drug: Dextromethorphan; Drug: Codeine; Drug: Morphine
- CYP2D6+ (Active Comparator): Extensive metabolizers (EM) of codeine
  Interventions: Drug: Dextromethorphan; Drug: Codeine; Drug: Morphine

INTERVENTIONS:
Drug: Dextromethorphan — one time dose - 0.3mg/kg PO
  Other Names: (+)-3-methoxy-17-methyl-9α,13α,14α-morphinan; DXM
Drug: Codeine — one time dose - 2mg/kg PO
  Other Names: 3-methylmorphine
Drug: Morphine — one time dose - 0.15mg/kg IV
  Other Names: MS Contin; MSIR

SUMMARY:
To develop and validate a non-invasive, in vivo, phenotyping method for CYP2D6 using the non-injurious neuroselective electrical stimulation technique: pain perception threshold/pain tolerance threshold (PPT/PTT) in children and adolescents with sickle cell disease.

DETAILED DESCRIPTION:
Codeine is a pro-drug with its analgesic activity being dependent on the metabolism of codeine to morphine. The metabolism of codeine to morphine is catalyzed by the cytochrome P450 enzyme 2D6 (CYP2D6) of which there are over 70 genetic variants leading to differing metabolic capabilities within populations. It is hypothesized that the changes in PPT/PTT will vary based on the individuals ability to convert morphine to codeine.

Ineffective analgesic management of patients with sickle cell disease remains a major problem in the management of the disorder in both adults and children. The pharmacological treatment of acute and chronic pain conditions resulting from vaso-occlusive crises in children with sickle cell disease typically involves the use of opioids. In the outpatient setting, this is most commonly achieved with administration of codeine and/or tramadol, both substrates of cytochrome P450 2D6 (CYP2D6). Currently these drugs are used in this patient population without any information concerning the patient's capacity to metabolize these CYP2D6 substrates which may lead to over and under treatment of pain depending on their CYP2D6 activity. The proposed objectives in this application will address this issue by the development of a pharmacodynamic assessment tool that will objectively assess the response to morphine in terms of analgesic response (pharmacodynamic assessment). This new tool might also serve as a non-invasive technique for CYP2D6 phenotyping if CYP2D6 substrates are used for pain therapy by assessing specifically morphine response. Development of this novel assessment tool will result in improved opioid analgesic therapy in this population. Future anticipated studies will examine the application of this technique in the determination of opioid tolerance and hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 7 to 18 years of age
* The subject is of African American descent
* The subject has sickle cell disease (HbSS)
* The subject has a history of vaso-occlusive crisis occurring within the 6 months prior to enrollment requiring opioid analgesia use
* The subject is willing to remain at the research site for the duration of each study session.
* The subject's parent / legal guardian has provided written informed consent to study participation
* The subject has provided written assent to study participation

Exclusion Criteria:

* The subject is a pregnant or lactation female (if post-menarchal, a negative pregnancy test must be confirmed on the day that any drug is administered (i.e., morphine, dextromethorphan or codeine)
* The subject has a history of smoking
* The subject has a history of alcohol use within the last 24 hours prior to testing session(s)
* The subject has a medical history of neuropathic pain, gastrointestinal, hepatic or renal disease
* The subject has a history of medication use including herbal therapies that are known to inhibit or induce CYP2D6 or morphine
* The subject has known or suspected hypersensitivities / allergies to codeine, morphine or dextromethorphan
* The subject is in active, vaso-occlusive crisis

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain Tolerance Threshold | 5 seconds
  5 measurements over 8 hours; 2 separate days

CONTACTS AND LOCATIONS:
Overall Officials: Julia C. Finkel, M.D., Principal Investigator — Children's National Medical Center-PPRU
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States